CLINICAL TRIAL: NCT03183271
Title: Phase II Clinical Study on Proton Therapy Boost (Hadrontherapy) for Locally Advanced HEAD AND NECK TUMORS
Brief Title: Proton Boost for Locally Advanced HEAD AND NECK TUMORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNAO 06/2011
Record Dates: First submitted 2017-06-04; First posted 2017-06-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Epithelial Tumor, Malignant; Neuroendocrine Tumors
MeSH Terms: conditions — Carcinoma; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: External beam radiotherapy (Experimental): A total of 20 patients will be irradiated with protons after photon IMRT
  Interventions: Radiation: external beam proton radiation therapy.

INTERVENTIONS:
Radiation: external beam proton radiation therapy. — Treatment of irradiation with protons beam The patients will be enrolled either at the Centro Nazionale di Adroterapia Oncologica (CNAO), Pavia, Italy, or at referral Hospitals enrolling head and neck patients for treatment with photon IMRT.

SUMMARY:
The aim of this research project is to test the local response and the acute toxicity (which can be observed within 90 days).

DETAILED DESCRIPTION:
Local response and acute toxicity are primary endpoints of the trial. At CNAO a proton boost is delivered on the PTV1rx (area at high risk of relapse) up to at least 70 Gy [RBE] in 2-3 Gy [RBE] per fractions for 8-15 total fractions.

PTV2 rx (area at low or intermediate risk of relapse) will be irradiated with photon IMRT up to a total dose of 50-60 Gy [RBE].

Secondary endpoints of the trial are local control, relapse free survival, overall survival, tumor specific survival, intermediate and long term toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologic/cytologic diagnosis of primary epithelial malignant or neuroendocrine tumour
* Inoperable tumour, locally advanced stage
* Seated in rhinopharynx, nasal and paranasal sinuses, hypopharynx, larynx, oral cavity and oropharynx
* At least one lesion measured according to the RECIST criteria
* Enrollment for irradiation with IMRT up to 50-60 Gy RBE] on the PTV1rx and PTV2 rx to be followed at CNAO with irradiation with proton boost on thePTV1rx.

Exclusion Criteria:

* Metastasis
* Previous radiotherapy
* Any metallic implants or other conditions such to prevent an adequate imaging of target volume
* Unavailability of previous IMRT first phase radiotherapy plans

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Local response | 90 days
  RECIST criteria
Acute toxicity | 90 days
  According to CTCAE v4.0

SECONDARY OUTCOMES:
Local control | 5 years
  RECIST criteria on MRI evaluation
Disease free survival | 5 years
  RECIST criteria on MRI evaluation - months from RT treatment to documented local relapse
Overall survival | 5 years
  On MRI and total body CT evaluation - months from RT treatment to death
Late toxicity | 5 years
  According to CTCAE v4.0 registered during follow up visits

CONTACTS AND LOCATIONS:
Locations (1):
- CNAO, Pavia, Italy